CLINICAL TRIAL: NCT07231809
Title: Hyperthermic Intravesical Chemotherapy (HIVEC) In Patients With BCG-Non Responsive Or Intolerant High-Grade BCG-Infiltrating Non-Muscle-Infiltrating Bladder Cancer And Not Eligible For Radical Cystectomy: Phase II Study (SMG-Bladder 01).
Brief Title: Hyperthermic Intravesical Chemotherapy (HIVEC) in BCG-Non-Responsive High-Grade NMIBC Patients
Acronym: HIVEC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AC.TA. S.r.l. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMG-Bladder 01
Record Dates: First submitted 2025-11-14; First posted 2025-11-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Non Muscle Invasive Bladder Cancer; Bladder Cancer; Carcinoma in Situ of Bladder; Urinary Bladder Neoplasms; Carcinoma, Transitional Cell, Bladder
Keywords: HIVEC; Hyperthermic Intravesical Chemotherapy; Mitomycin C; BRS Combat System; Bladder Tumor Recurrence; High-Grade Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms; Carcinoma

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, non-randomized, Phase II therapeutic study evaluating hyperthermic intravesical chemotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIVEC Treatment Arm (Experimental): Participants will receive Hyperthermic Intravesical Chemotherapy (HIVEC) with Mitomycin C according to the study protocol (induction + maintenance schedule). Mitomycin C is an approved medicinal product used within routine clinical practice. HIVEC is performed using a CE-marked recirculation system that maintains the solution at a controlled therapeutic temperature.
  Interventions: Procedure: Hyperthermic Intravesical Chemotherapy (HIVEC)

INTERVENTIONS:
Procedure: Hyperthermic Intravesical Chemotherapy (HIVEC) — Intravesical administration of Mitomycin C heated to approximately 43°C using a CE-marked recirculation system (BRS Combat device). Mitomycin C is supplied by the treating hospital as part of routine clinical practice. The procedure consists of 6 weekly instillations followed by 9 monthly instillations.
  Other Names: HIVEC System; BRS Combat

SUMMARY:
This is a Phase II, prospective, single-arm, open-label clinical study evaluating hyperthermic intravesical chemotherapy (HIVEC) with Mitomycin C in patients with high-grade, non-muscle-invasive bladder cancer (NMIBC) who are BCG-non-responsive or BCG-intolerant and are ineligible for, or refuse, radical cystectomy. Mitomycin C is an approved medicinal product used within routine clinical practice and administered with a CE-marked recirculation device (BRS Combat system) that maintains the solution at approximately 43°C for 60 minutes. The treatment schedule consists of 6 weekly induction instillations followed by 9 monthly maintenance instillations.

The co-primary objectives are to describe the safety and toxicity profile of HIVEC, including treatment discontinuations due to procedure-related toxicity, and to estimate the 12-month recurrence-free survival (12moRFS). Secondary objectives include characterizing patterns of non-muscle-invasive and muscle-invasive recurrences, bladder cancer-specific survival, overall survival, and quality of life. Approximately 50 patients will be enrolled in this single-center pilot study to generate exploratory safety and efficacy data in this high-risk population and to support the design of future randomized trials

DETAILED DESCRIPTION:
This is an interventional, prospective, single-center, single-arm, open-label, Phase II study conducted in patients with high-grade non-muscle-invasive urothelial carcinoma of the bladder (NMIBC) who are BCG-non-responsive or BCG-intolerant according to European Association of Urology criteria, and who are either not eligible for, or decline, radical cystectomy. Radical cystectomy remains the standard of care in this setting, but many patients are unfit because of age or comorbidities or are unwilling to undergo major surgery. Hyperthermic intravesical chemotherapy (HIVEC) has emerged as a potential alternative option for disease control in these high-risk patients. ￼

In this study, Mitomycin C 40 mg in 40 mL of sterile water is administered intravesically using the CE-marked BRS Combat recirculation system, which keeps the solution at a controlled temperature of about 43°C for 60 minutes. The treatment regimen includes an induction phase of 6 weekly instillations followed by a maintenance phase of 9 monthly instillations. Therapy may be discontinued earlier in the event of disease progression or unacceptable toxicity. Mitomycin C is purchased by the ASL Napoli 2 Nord as part of routine care, with costs reimbursed by the sponsor, while the device and related disposables are supplied on loan for use for the study. ￼

The co-primary endpoints are: (1) toxicity and safety, including the type, incidence, severity, and timing of adverse events graded according to NCI CTCAE v5.0 and PRO-CTCAE, and the proportion of patients who discontinue treatment due to procedure-related toxicity; and (2) 12-month recurrence-free survival (12moRFS), defined as the time from first instillation to recurrence or progression (Ta, T1, or CIS) or death from any cause, with estimates obtained using the Kaplan-Meier method. Secondary endpoints include the rate of Ta-T1 non-muscle-invasive recurrences, the proportion of muscle-invasive recurrences (≥T2), bladder cancer-specific survival, overall survival, and quality of life assessed with the EORTC QLQ-NMIBC24 questionnaire at predefined time points during treatment and follow-up. ￼

Approximately 50 patients will be enrolled between November 2025 and November 2026 at the Oncology and Urology Units of the "S. Maria delle Grazie" Hospital in Pozzuoli (ASL Napoli 2 Nord). Data will be recorded in an electronic database using anonymized patient codes. Statistical analyses will be primarily descriptive and exploratory, reflecting the monocentric, non-comparative design and the pilot nature of the study, with the aim of characterizing the safety profile of HIVEC and providing a preliminary estimate of 12-month recurrence-free survival and overall disease control in this population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Histologically confirmed high-grade non-muscle-invasive bladder cancer (NMIBC), including Ta, T1, and/or carcinoma in situ (CIS).
* BCG-unresponsive or BCG-intolerant disease according to international definitions (persistent or recurrent high-grade NMIBC after adequate BCG therapy).
* Patient is ineligible for, or refuses, radical cystectomy.
* Candidate for hyperthermic intravesical chemotherapy (HIVEC) according to clinical judgment.
* ECOG Performance Status 0-2.
* Adequate organ function according to institutional standards.
* Ability and willingness to comply with study procedures and follow-up schedule.
* Written informed consent obtained.

Exclusion Criteria:

* Muscle-invasive bladder cancer (≥ T2) or metastatic disease.
* Active urinary tract infection at baseline.
* Previous treatment with HIVEC or other intravesical hyperthermia systems.
* Known hypersensitivity to Mitomycin C or contraindications to intravesical chemotherapy.
* Active uncontrolled bleeding or gross hematuria preventing intravesical instillation.
* Upper urinary tract urothelial carcinoma.
* Pregnant or breastfeeding women.
* Any medical or psychological condition that, in the investigator's judgment, could interfere with study participation or compromise patient safety.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Treatment-Related Adverse Events (AEs) | Up to 12 months
  Incidence, type, timing, and severity of adverse events graded according to NCI CTCAE v5.0. Includes local and systemic toxicities related to hyperthermic intravesical chemotherapy and the proportion of patients who discontinue treatment due to toxicity.
12-Month Recurrence-Free Survival (RFS) | 12 months after completion of the HIVEC treatment schedule
  Proportion of patients who remain free from histologically confirmed recurrence of non-muscle-invasive bladder cancer (Ta, T1, or CIS) at 12 months from initiation of HIVEC treatment. Recurrence is defined per standard cystoscopic and histological criteria.

SECONDARY OUTCOMES:
Rate of non-muscle-invasive (Ta-T1) bladder cancer recurrences | Up to 12 months
  Percentage of patients experiencing a histologically confirmed Ta or T1 recurrence during the 12-month follow-up period.
Rate of muscle-invasive (≥T2) recurrences | Up to 12 months
  Percentage of patients who progress to muscle-invasive bladder cancer (≥T2) confirmed by imaging or histology.
Cancer-specific survival | up to 12 months
  Assessing cancer-specific survival (bladder)
Overall Survival (OS) | Up to 12 months
  Time from first HIVEC instillation to death from any cause.
Quality of Life (QoL) | Up to 12 months
  Quality of life will be assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire - Non-Muscle-Invasive Bladder Cancer Module (EORTC QLQ-NMIBC24).
  The questionnaire generates multi-item symptom and function scales scored from 0 to 100, where higher scores indicate worse symptoms or lower functioning in accordance with the official EORTC scoring manual

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Facchini, MD, Principal Investigator — P.O. "Santa Maria delle Grazie" - ASL Napoli 2 Nord
Locations (1):
- P.O. "Santa Maria delle Grazie" - ASL Napoli 2 Nord, Pozzuoli, Italy

IPD SHARING:
Plan to Share IPD: Undecided
The decision regarding IPD sharing is not finalized. Potential data sharing will depend on institutional policies, GDPR requirements, and Ethics Committee approval. Any sharing would involve only de-identified data and would require a formal data sharing agreement.